CLINICAL TRIAL: NCT05762354
Title: Investigation of the Relationship Between Body Image Perception, Proprioception, Cobb Angle and Posture in Individuals With Adolescent Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Istanbul Gelisim University (Other)
Responsible Party: Principal Investigator, Aysem Ecem Ozdemir, Research Assistant, Istanbul Gelisim University
Other Study IDs: GUS001
Record Dates: First submitted 2023-02-28; First posted 2023-03-09 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Scoliosis; Adolescence; Scoliosis Idiopathic
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Scoliosis Group: Adolescent Idıopathic Scoliosis

SUMMARY:
Scoliosis is a three-dimensional torsional deformation of the spine and trunk. Chest deformity and pelvic asymmetry are often seen together with spinal deformity. Adolescent idiopathic scoliosis occurs from the onset of puberty until growth plate closure and is the most common of all scoliosis. One of the most common deformities among posture disorders is known as scoliosis. The change in load distribution resulting from this three-dimensional deformation causes postural changes in patients with idiopathic scoliosis. According to a study, it is thought that postural control and central information processing efficiency may decrease as the Cobb angle increases in people with scoliosis.

DETAILED DESCRIPTION:
Scoliosis, shoulder asymmetry, midline asymmetry, trunk shift and lower extremity length inequality. Therefore, it affects body image perception negatively by limiting physical functions and mobility. In a study conducted with individuals with AIS, it was found that as the Cobb angle increased, body image was adversely affected.

It is also known that during the vertebral growth period in idiopathic scoliosis, postural reflex mechanisms originating from the proprioceptive organs and balance problems are associated with the displacement of the vertebrae. As a result of a study on vestibular effect and proprioception, it is concluded that it would be beneficial to include proprioception, balance and coordination exercises in the treatment of scoliosis. In the current literature review, no study was found that investigated the relationships between Cobb angle, proprioception, body image perception and posture variables in individuals with Adolescent Idiopathic Scoliosis.

The aim of our study is to explain the relationship between some problems accompanied by scoliosis in individuals diagnosed with idiopathic scoliosis. With the results that can be obtained from our study, we aim to explain how posture, proprioception and body image perception are affected in individuals with AIS and to contribute to the exercise programs that can be given to the person in line with these results.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with adolescent idiopathic scoliosis by a doctor,
* Not having cognitive, mental and psychological problems,
* Continuing exercise or brace therapy.

Exclusion Criteria:

* Having a history of spinal surgery
* Having a type of scoliosis other than idiopathic,
* Presence of musculoskeletal system pathologies,
* Vestibular system disorders.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents Idıopatic Scoliosis
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Fukuda Step Test | Baseline
  The patient will do a 50 or 100 step counting motion with eyes open and closed. 30 degree rotation or 50 cm displacement for 50 steps relative to the starting position; For 100 steps, 31 turns of 45 degrees and displacement of 100 cm will count as a positive result. The hypoactive side of the labyrinth will be accepted as the patient's turning side. The displacement amount of the person will be measured in cm with the help of a tape measure, and the rotation amount will be measured in degrees with the help of a goniometer and recorded in the evaluation form.

SECONDARY OUTCOMES:
Cobb Degree | Baseline
  It can be measured with the help of a goniometer or digitally as the angle between the lines perpendicular to the parallels drawn on the corpus of the first and last vertebrae participating in the curvature. The 'Cobb' angle is the gold standard in the evaluation of scoliosis.
Trunk Rotation | Baseline
  In the study, evaluations with scoliometer will be performed standing and sitting, in the forward bending position until the trunk is in a horizontal position and the scapula and pelvis are aligned. Vertebral rotation angle values taken from the thoracic, thoracolumbar and lumbar regions will be measured by the training physiotherapist and the highest angular value will be recorded as ATR.
Posterior Trunk Symmetry Index | Baseline
  The POTSI parameter is defined as the sum of six indices: the frontal plane asymmetry index (C7, axilla folds and waist lines) and the three frontal plane height difference indexes (acromions, axilla folds, and waist lines). The POTSI score is calculated by placing the indices on the photograph of the patient transplanted from the posterior.
Walter Reed Visual Assessment Scale | Baseline
  In addition to understanding the visual change caused by scoliosis, the scale used to evaluate the treatment results evaluates the deformity under 7 headings. These; spine curvature, rib protrusion, lumbar protrusion, thorax deformity relative to pelvis, trunk imbalance, shoulder and scapula asymmetry. Each of the domains is scored from 1 to 5 with worsening deformity for increasing scores.
SRS 22 Questionaire | Baseline
  SRS-22 is the most commonly used questionnaire to evaluate quality of life in scoliosis patients. The questionnaire is a simple and practical quality of life questionnaire, which has been translated into our language and has validity and reliability, created specifically for individuals with scoliosis. Each question is scored from 1 (worst) to 5 (best) in the questionnaire, which assesses five domains: function, pain, self-image, mental health (five questions each), and treatment satisfaction (two questions).
Coronal Imbalance | Baseline
  In the frontal plan evaluation, the plumb line is suspended in line with the midline of the sacrum, the deviation from the midline at the C7 level is measured and recorded in the evaluation form in cm. clinical threshold for plumb line distances; It will be 50 mm for C7 and 60 mm for L3.
Sagittal Index | Baseline
  In order to detect deformities that develop different from the neutral, by hanging the pendulum from the point where the dorsal kyphosis is most prominent in the sagittal plane; At C7, T12 and L3 alignments, the distance from the pendulum to the spinous process is measured in cm and will be recorded on the evaluation form. If a value greater than 90 mm is obtained as a result of the sagittal index, which is the sum of C7 and L3, it is accepted that the score obtained is correlated with increased kyphosis.

CONTACTS AND LOCATIONS:
Overall Officials: İrem Kurt, Msc., Principal Investigator — İstanbul Gelişim Üniversitesi
Locations (1):
- İstanbul Gelişim Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided